CLINICAL TRIAL: NCT02775994
Title: Ilaris (Canakinumab) in Patient With Periodic Fever, Aphthous Stomatitis, Pharyngitis and Cervical Adenitis (PFAPA)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0032-16-RMC
Record Dates: First submitted 2016-04-27; First posted 2016-05-18 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Periodic Fever
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Single dose of Canakinumab 4mg/kg
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — interleukin beta (IL-1) antagonist
  Other Names: Ilaris

SUMMARY:
Periodic Fever, Aphthous stomatitis, Pharyngitis and cervical Adenitis (PFAPA) is one of the most common, least explored periodic fever syndrome in childhood. This study aims to investigate whether a single dose of an interleukin beta (IL-1) antagonist, Canakinumab will be able to abort PFAPA flares in patients who experience a flare in an average of 2 weeks or less. This will be a single arm open label pilot study. 10 patients will be recruited from 1 center (Pediatric rheumatology unit -Schneider children's medical center of Israel).

Patients in ages 2-10 years old who are diagnosed with PFAPA according to clinical criteria at least 3 months prior to enrollment and who are under regular care for this disease (single dose of glucocorticoids during flare) and who suffer from more than 4 PFAPA flares for the last 2 months, will be screened for this study. In the second documented flare, patients will be enrolled to receive a single dose of subcutaneous (SC) Canakinumab 4 mg/kg. The primary outcome is defined as - 50% reduction in PFAPA flares for the next 2 consecutive months as reported by the patient (use of diary) and documented by the patient primary care physician and/ or the researcher in a monthly follow up visits. Secondary outcome measure are define as time to flare (days) and Parent/patient quality of life assessment measured by 100mm visual analog scale (VAS).

DETAILED DESCRIPTION:
Study Objectives:

Primary objective: Patients will experience at least 50% reduction in PFAPA flares for the next 2 consecutive months after receiving single dose of canakinumab (4 mg/kg).

Secondary objectives:

1. Time to flare
2. Parent/patient quality of life assessment

Study rationale:

Periodic Fever, Aphthous stomatitis, Pharyngitis and cervical Adenitis (PFAPA) is one of the most common, least explored periodic fever syndrome in childhood. It was discovered only in 1987 by Marshall et al. who noticed periodic attacks of fever along with pharyngitis and cervical adenitis mimicking streptococcal acute tonsillitis. Many of these patients were erroneously treated with antibiotic despite negative throat cultures. The exact prevalence of this syndrome is not known but PFAPA seems to be far more frequent than other auto-inflammatory diseases . Since PFAPA has an unknown etiology and lacks a specific laboratory marker, the diagnosis is made by using clinical criteria which include more than three documented episodes of fever, lasting no more than five days and occurring at regular intervals at a range of three to six weeks, pharyngitis plus tender cervical lymphadenopathy or aphthous ulcers, normal growth parameters and good health between episodes . Single dose of glucocorticoids usually leads to prompt resolution of the disease. Their usefulness as therapy, however, is limited by the fact that glucocorticoid treatment results in shortening the interval between attacks in about 30 percent of case up to even weekly attacks. Prophylaxis therapy with cimetidine or colchicine has limited value and most children do not respond. Some physicians will try to use them, mainly in patients who suffer from frequent attacks despite glucocorticoids therapy as the last resort before tonsillectomy, however, many children eventually will undergo tonsillectomy which, in many cases, does not prevent the attacks and may cause morbidity and even mortality. The pathogenesis of PFAPA is still not fully understood. However, the rapid response to corticosteroid treatment suggests an immune dysregulation. Recent studies suggest, as in other autoinflammatory syndromes, an essential role of the innate immune system by activation of the inflammasome during fever attacks which leads to production of Interleukin 1 along with other proinflammatory cytokines and chemokines and indeed, treatment with anakinra has been reported to cause remission in an adult patient with resistant PFAPA and is in clinical use in several medical centers in the US.

Timelines and Study duration:

Start date: within 2 months after Helsinki committee approval- estimated first patient first visit (FPFV) -1 month Estimated Last Patient Last treatment (LPLT) last patient first treatment (LPFT)/last patient (LP) enrollment - 6 months End date: 6 months after last patient enrollment Once enrolled, patients will receive a single dose of Canakinumab and then will be followed for a period of a total 24 weeks after receiving Canakinumab - weekly during the first month and then monthly for the next 5 months.

Study Report date: within 4 month after Last Patient Last Visit. Publication date: within 10 month after Last Patient Last Visit.

Methodology:

This will be a single arm open label pilot study. This study will be approved by our institutional and national Helsinki committees. Patients in ages 2-10 years old who are diagnosed with PFAPA according to clinical criteria at least 3 months prior to enrollment and who are under regular care for this disease (single dose of glucocorticoids during flare) and who suffer from more than 4 PFAPA flares for the last 2 months, will be screened for this study. Patients with another chronic disease, neutropenia, elevated liver enzymes or in which the diagnosis of PFAPA is in doubt, will be excluded. In addition patients that receive treatment with cimetidine/famotidine, montelukast or colchicine will undergo a washout period of 2 weeks (see appendix).

. Screening period: After signing the informed consent and filling demographic and clinical questionnaires, the patient will enter a screening period of one month. At the screening visit, participants will undergo purified protein derivative (PPD) test to rule out tuberculosis and laboratory workup which includes: Complete blood count (CBC), full chemistry panel, erythrocyte sedimentation rate (ESR), C reactive protein (CRP) and urinalysis. During this period, the first PFAPA flare will be treated with a single dose of oral glucocorticoids (which is given as part of their regular care) and the response will be documented by the PI or co-PI in a formal study visit.

Enrolment: In the second documented flare, patients will be enrolled to receive a single dose of SC Canakinumab 4 mg/kg. Treatment with glucocorticoids during the second flare will not be allowed.

Patients who have less than 2 flares during the screening period will have the option to be enrolled in the next consecutive month as long as they have 2 documented PFAPA flares at that month. Patients, who fail to flare in that phase as well, will be censored (screening failure).

Once a patient experiences a flare after the administration of canakinumab, He will be treated according to the clinician/ researcher decision (e.g. - a dose of corticosteroids). All flares will be documented during the follow-up period.

Number of centers & patients: 10 patients will be recruited from 1 center (Pediatric rheumatology unit -Schneider children's medical center of Israel). Potential patients from other pediatric rheumatology clinics around the country will be referred to our clinic.

Sample size justification: This is a pilot study and it is not powered for statistical significance.

Population:

Key inclusion criteria

1. Patients in ages 2-10 years old who are diagnosed with PFAPA at least 3 months prior to enrollment according to clinical criteria will be screened for this study.
2. Suffer from more than 4 PFAPA flares 2 months prior to the screening period.
3. Have signed informed consent for the study.
4. Have at least 2 documented PFAPA flare during the screening period.

Key exclusion criteria

1. Patients who are diagnosed with chronic disease including another auto inflammatory disease.
2. Patients who suffer from neutropenia or elevated liver enzymes.
3. Patients who receive treatment with cimetidine/famotidine, montelukast or colchicine 2 weeks or less prior to enrollment.

Pharmacovigilance requirements:

Definition of an AE: Any untoward medical occurrence in a subject administered a pharmaceutical product that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the investigational medicinal product.

Investigational Medicinal Product (IMP) includes the drug under evaluation and the comparator drug(s) if specified as part of the research objective, given at any time during the study. Medical conditions/diseases present before starting the drug of interest are only considered adverse events if they worsen after starting the drug of interest.

The occurrence of adverse events will be sought by non-directive questioning of the patient at each visit during the study. Adverse events also may be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments. All adverse events will be recorded in the study database including the following information:

1. severity grade (mild, moderate, severe)
2. its relationship to the drug(s) of interest (suspected/not suspected)
3. its duration (start and end dates or if continuing at final exam)
4. whether it constitutes a serious adverse event (SAE)

A SAE is any untoward medical occurrence that at any dose:

* results in death,
* is life-threatening,
* requires inpatient hospitalization or prolongation of existing hospitalization,
* results in persistent or significant disability/incapacity,
* is a congenital anomaly/birth defect,
* is otherwise a significant medical event. This includes any SAEs likely to arise from the trial indication or progression of underlying/concomitant illness (e.g. progression of cancer in oncology trials), unless specified in the protocol as study specific exemptions.

Any SAE, irrespective of causality, occurring after the subject has provided informed consent and until four weeks after the subject has stopped study participation must be reported unless otherwise stated in the protocol. SAEs occurring after four weeks from ending study participation should only be reported if considered by the Investigator attributable to the exposure to the investigational drug(s) during the trial period. This includes the period in which the study protocol interferes with the standard medical treatment given to a subject, even if study treatment has not yet started (e.g. withdrawal of previous treatment during washout period, change in treatment to a fixed dose of concomitant medication).

Timelines: All serious adverse events (SAEs) from interventional clinical trials must be reported by the sites to Sponsor within 24 hours of occurrence of the SAE. The timelines for investigator initiated trials reporting to Novartis will be done as per Third Party Study/Investigator Initiated Trial Agreement.

Follow-up reports:

SAEs will be followed until resolution or until it is judged to be permanent, and an assessment will be made at each visit (or more frequently, if necessary) of any changes in severity, the suspected relationship to the drug of interest, the interventions required to treat it, and the outcome.

The Sponsor shall support Novartis in the following-up of all SAEs so that complete information is available to maintain patient safety and also as part of any commitments by Novartis to any Health authority OR specific Health authority follow-up requests for the product under investigation.

Pregnancies: N/A

Evaluation criteria:

Primary endpoint:

Efficacy measure - 50% reduction in PFAPA flares for the next 2 consecutive months as reported by the patient (use of diary) and documented by the patient primary care physician and/ or the researcher in a monthly follow up visits. This will be compared to the average number of flares (per 2 months) during the last 3 consecutive months before therapy (i.e number of flares in last 3 months before therapy divided by 3 and multiplied by 2).

Secondary endpoints:

1. Time to flare (period between administration of a single dose of canakinumab until the first documented PFAPA flare. Will be compared to the average time between 2 consecutive flares before therapy (e.g.: first documented flare- will be day 1. In the following 90 days 5 more flares ( 3 before screening and 2 after)= 90/5= 18d mean time to flare).
2. Parent/patient quality of life assessment measured by 100mm visual analog scale (VAS) difference at screening vs. 2 months after administration of a single dose of canakinumab.

ELIGIBILITY:
Key inclusion criteria

1. Patients in ages 2-10 years old who are diagnosed with PFAPA at least 3 months prior to enrollment according to clinical criteria will be screened for this study.
2. Suffer from more than 4 PFAPA flares 2 months prior to the screening period.
3. Have signed informed consent for the study.
4. Have at least 2 documented PFAPA flare during the screening period.

Key exclusion criteria

1. Patients who are diagnosed with chronic disease including another auto inflammatory disease.
2. Patients who suffer from neutropenia or elevated liver enzymes.
3. Patients who receive treatment with cimetidine/famotidine, montelukast or colchicine 2 weeks or less prior to enrollment.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in average number of flares - documented by the use of diary | baseline (canakinumab administration) and 2 months after baseline
  Efficacy measure - 50% reduction in PFAPA flares for the next 2 consecutive months as reported by the patient (use of diary) and documented by the patient primary care physician and/ or the researcher in a monthly follow up visits. This will be compared to the average number of flares (per 2 months) during the last 3 consecutive months before therapy (i.e number of flares in last 3 months before therapy divided by 3 and multiplied by 2).

SECONDARY OUTCOMES:
Time to flare - documented by the use of diary | baseline (canakinumab administration) and up to 24 weeks after baseline
  Time to flare - period between administration of a single dose of canakinumab until the first documented PFAPA flare as reported by the patient (use of diary) and documented by the patient primary care physician and/ or the researcher in a monthly follow up visits. Will be compared to the average time between 2 consecutive flares before therapy (e.g: first documented flare- will be day 1. In the following 90 days 5 more flares (3 before screening and 2 after) = 90/5= 18d mean time to flare).
Change in quality of life - documented by the use of questionnaire | at the time of screening visit and 2 months after baseline (canakinumab administration)
  Parent/patient quality of life assessment measured by 100mm visual analog scale (VAS) difference at screening vs. 2 months after administration of a single dose of canakinumab.

CONTACTS AND LOCATIONS:
Overall Officials: Liora Harel, MD, Principal Investigator — SCMCI
Locations (1):
- SCMCI, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided